CLINICAL TRIAL: NCT06219031
Title: A Study of the Tumor Microenvironment Affecting the Efficacy of Immunotherapy for Esophageal Cancer
Status: Completed | Type: Observational
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Principal Investigator, Yongshun Chen, professor, Renmin Hospital of Wuhan University
Other Study IDs: WDRY2024-K007
Record Dates: First submitted 2024-01-12; First posted 2024-01-23 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — FFPE
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- valid group（CR/PR）: CR/PR
  Interventions: Other: no intervention
- invalid group（SD/PD）: SD/PD
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
This study is a retrospective study of clinical specimens. The study subjects were patients with esophageal cancer who received immunotherapy. Tumor tissue specimens surgically removed from patients before treatment will be collected primarily. In situ immunohistochemistry and multicolor immunofluorescence will be performed. We hypothesize that there are differences in lipid metabolism-related proteins in tumor tissues and immune cells in the preexisting tumor microenvironment in patients with esophageal cancer prior to immunotherapy, and that there is a link between such differences and the efficacy of immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Esophageal cancer patients receiving immunotherapy
2. Radical esophagectomy for esophageal cancer at our institution prior to receiving immunotherapy
3. Age greater than or equal to 18 years and less than or equal to 75 years old Imaging to assess patient efficacy after cycle 2 immunotherapy (CR/PR, SD/PD according to recist 1.1)
4. Pathology Tumor tissue available

Exclusion Criteria:

1. Clinical and pathologic information not available
2. Combined history of other malignant tumors
3. Unavailability of surgically resected tissue
4. Preoperative neoadjuvant therapy
5. Radical esophagectomy for esophageal cancer not performed prior to immunotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with esophageal cancer receiving immunotherapy
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Immunotherapy efficacy | 2018-2022
  Imaging to assess patient efficacy after cycle 2 immunotherapy (CR/PR, SD/PD according to Recist 1.1)
CR、PR、SD、PD | 2018-2022
  CR：All target lesions disappear and the short diameter of all pathologic lymph nodes (both target and non-target nodes) must be reduced to <10 mm.
  PR：At least 30% reduction in the sum of target lesion diameters from baseline levels SD：A relative increase in diameter sum of at least 20% (or the baseline value if the baseline measurement is minimal), referenced to the minimum of the sum of the diameters of all measured target lesions throughout the course of the experimental study; in addition to this, an increase in the absolute value of diameter sum of at least 5 mm must be met (the presence of one or more new lesions is also considered to be disease progression).
  Translated with www.DeepL.com/Translator (free version) PD：The target lesion did not decrease to the level of PR, nor did it increase to the level of PD, and in between, the minimum value of the sum of the diameters can be used as a reference for the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Renmin hosptial of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Result] Fang P, Zhou J, Liang Z, Yang Y, Luan S, Xiao X, Li X, Zhang H, Shang Q, Zeng X, Yuan Y. Immunotherapy resistance in esophageal cancer: Possible mechanisms and clinical implications. Front Immunol. 2022 Sep 2;13:975986. doi: 10.3389/fimmu.2022.975986. eCollection 2022. PMID 36119033
- [Result] Li Q, Liu T, Ding Z. Neoadjuvant immunotherapy for resectable esophageal cancer: A review. Front Immunol. 2022 Dec 8;13:1051841. doi: 10.3389/fimmu.2022.1051841. eCollection 2022. PMID 36569908
- [Result] Lei X, Lei Y, Li JK, Du WX, Li RG, Yang J, Li J, Li F, Tan HB. Immune cells within the tumor microenvironment: Biological functions and roles in cancer immunotherapy. Cancer Lett. 2020 Feb 1;470:126-133. doi: 10.1016/j.canlet.2019.11.009. Epub 2019 Nov 12. PMID 31730903
- [Result] Yin J, Yuan J, Li Y, Fang Y, Wang R, Jiao H, Tang H, Zhang S, Lin S, Su F, Gu J, Jiang T, Lin D, Huang Z, Du C, Wu K, Tan L, Zhou Q. Neoadjuvant adebrelimab in locally advanced resectable esophageal squamous cell carcinoma: a phase 1b trial. Nat Med. 2023 Aug;29(8):2068-2078. doi: 10.1038/s41591-023-02469-3. Epub 2023 Jul 24. PMID 37488287
- [Result] Arbore G, Albarello L, Bucci G, Punta M, Cossu A, Fanti L, Maurizio A, Di Mauro F, Bilello V, Arrigoni G, Bonfiglio S, Biancolini D, Puccetti F, Elmore U, Vago L, Cascinu S, Tonon G, Rosati R, Casorati G, Dellabona P. Preexisting Immunity Drives the Response to Neoadjuvant Chemotherapy in Esophageal Adenocarcinoma. Cancer Res. 2023 Sep 1;83(17):2873-2888. doi: 10.1158/0008-5472.CAN-23-0356. PMID 37350667
- [Result] Parra ER, Zhang J, Jiang M, Tamegnon A, Pandurengan RK, Behrens C, Solis L, Haymaker C, Heymach JV, Moran C, Lee JJ, Gibbons D, Wistuba II. Immune cellular patterns of distribution affect outcomes of patients with non-small cell lung cancer. Nat Commun. 2023 Apr 25;14(1):2364. doi: 10.1038/s41467-023-37905-y. PMID 37185575
- [Result] Koundouros N, Poulogiannis G. Reprogramming of fatty acid metabolism in cancer. Br J Cancer. 2020 Jan;122(1):4-22. doi: 10.1038/s41416-019-0650-z. Epub 2019 Dec 10. PMID 31819192
- [Result] Ma X, Bi E, Lu Y, Su P, Huang C, Liu L, Wang Q, Yang M, Kalady MF, Qian J, Zhang A, Gupte AA, Hamilton DJ, Zheng C, Yi Q. Cholesterol Induces CD8+ T Cell Exhaustion in the Tumor Microenvironment. Cell Metab. 2019 Jul 2;30(1):143-156.e5. doi: 10.1016/j.cmet.2019.04.002. Epub 2019 Apr 25. PMID 31031094
- [Result] Yang W, Bai Y, Xiong Y, Zhang J, Chen S, Zheng X, Meng X, Li L, Wang J, Xu C, Yan C, Wang L, Chang CC, Chang TY, Zhang T, Zhou P, Song BL, Liu W, Sun SC, Liu X, Li BL, Xu C. Potentiating the antitumour response of CD8(+) T cells by modulating cholesterol metabolism. Nature. 2016 Mar 31;531(7596):651-5. doi: 10.1038/nature17412. Epub 2016 Mar 16. PMID 26982734
- [Result] Su P, Wang Q, Bi E, Ma X, Liu L, Yang M, Qian J, Yi Q. Enhanced Lipid Accumulation and Metabolism Are Required for the Differentiation and Activation of Tumor-Associated Macrophages. Cancer Res. 2020 Apr 1;80(7):1438-1450. doi: 10.1158/0008-5472.CAN-19-2994. Epub 2020 Feb 3. PMID 32015091
- [Result] Lim SA, Wei J, Nguyen TM, Shi H, Su W, Palacios G, Dhungana Y, Chapman NM, Long L, Saravia J, Vogel P, Chi H. Lipid signalling enforces functional specialization of Treg cells in tumours. Nature. 2021 Mar;591(7849):306-311. doi: 10.1038/s41586-021-03235-6. Epub 2021 Feb 24. PMID 33627871
- [Result] Xu C, Sun S, Johnson T, Qi R, Zhang S, Zhang J, Yang K. The glutathione peroxidase Gpx4 prevents lipid peroxidation and ferroptosis to sustain Treg cell activation and suppression of antitumor immunity. Cell Rep. 2021 Jun 15;35(11):109235. doi: 10.1016/j.celrep.2021.109235. PMID 34133924
- [Result] Gao L, Chen Y. A metabolomic and proteomic study to elucidate the molecular mechanisms of immunotherapy resistance in patients with oesophageal squamous cell carcinoma. Biomed Rep. 2023 Apr 6;18(5):36. doi: 10.3892/br.2023.1619. eCollection 2023 May. PMID 37089578